CLINICAL TRIAL: NCT02054481
Title: A 48 Weeks Study of Three Different Dose Regimens of BI 655066 Administered Subcutaneously in Patients With Moderate to Severe Chronic Plaque Psoriasis (Randomised, Dose-ranging, Active-comparator-controlled (Ustekinumab), Double-blind Within Dose Groups of BI 655066)
Brief Title: BI 655066 Dose Ranging in Psoriasis, Active Comparator Ustekinumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1311.2; 2012-004384-48 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; Ustekinumab

ARMS (4):
- Arm 1 (Experimental): BI 655066 s.c.
  Interventions: Drug: BI 655066
- Arm 2 (Experimental): BI 655066 s.c.
  Interventions: Drug: BI 655066
- Arm 3 (Experimental): BI 655066 s.c.
  Interventions: Drug: BI 655066
- Arm 4 (Active Comparator): Ustekinumab s.c.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: BI 655066 — Medium dose
  Arms: Arm 2
Drug: BI 655066 — High dose
  Arms: Arm 3
Drug: Ustekinumab
  Arms: Arm 4
Drug: BI 655066 — Low dose
  Arms: Arm 1

SUMMARY:
The overall purpose of this trial is to assess clinical efficacy and safety of different subcutaneous doses of BI 655066 in adult patients with chronic plaque psoriasis in order to select doses for further clinical trials.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index (BMI) >/= 18.5 and < 40 kg/m²
* Patients with stable moderate to severe chronic plaque-type psoriasis with or without psoriatic arthritis involving >/= 10% body surface area, with disease severity PASI >/= 12 and sPGA score of moderate and above (score of at least 3) at screening visit and visit 2 (randomisation), as assessed by the investigator
* Psoriasis disease duration of at least 6 months prior to screening, as assessed by the investigator
* Patients must be candidates for systemic psoriasis treatment or phototherapy, as assessed by the investigator
* Patients must be suitable candidates for ustekinumab (Stelara®) therapy as given in the local labelling
* Patient must give informed consent and sign an approved consent form prior to any study procedures in accordance with GCP and local legislation

Exclusion criteria:

* Patients with guttate, erythrodermic, or pustular psoriasis and patients with drug-induced psoriasis, as diagnosed by the investigator
* Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and ECG), that in the opinion of the investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied. (Psoriatic arthritis is not considered an exclusion criterion)
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders, or history of orthostatic hypotension, fainting spells or blackouts, that in the investigator's judgement, could jeopardize the safe conduct of the study.
* Clinically important acute or chronic infections including hepatitis and HIV.

With regards to tuberculosis the following applies:

Have signs or symptoms suggestive of current active or latent TB upon medical history, physical examination and/or a chest radiograph (both posterior-anterior and lateral views, taken within 3 months prior to the first administration of study drug and read by a qualified radiologist).

Have history of latent or active TB prior to screening, except for patients who have documentation of having completed an adequate treatment regimen at least 6 months prior to the first administration of study agent.

Have positive IGRA testing (QuantiFERON-TB Gold) within 2 months prior to or during screening, in which active TB has not been ruled out, except for patients with history of latent TB and documentation of having completed an adequate treatment regimen at least 6 months prior to the first administration of study agent.

* Have had a live vaccination </= 12 weeks prior to randomisation (visit 2). Patients must agree not to receive a live vaccination during the study. No BCG vaccines should be given for one year prior to randomisation (visit 2), during the study and for one year after last administration of study drug (according to the Stelara® SPC).
* History of clinically significant hypersensitivity to a systemically administered biologic agent or its excipients
* History of malignancy in the past 5 years or suspicion of active malignant disease except treated cutaneous squamous cell or basal cell carcinoma
* Has received any therapeutic agent directly targeted to IL-12, IL-23 (including ustekinumab (Stelara®))
* Use of biologic agents within 12 weeks (infliximab, etanercept, adalimumab, other biologics) prior to treatment, systemic anti-psoriatic medications or phototherapy within 4 weeks prior to treatment, or topical anti-psoriasis medications within 2 weeks prior to treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (32):
- United States (12):
  - 1311.2.10010 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1311.2.10013 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1311.2.10003 Boehringer Ingelheim Investigational Site, Arlington Hts, Illinois
  - 1311.2.10002 Boehringer Ingelheim Investigational Site, Bay City, Michigan
  - 1311.2.10004 Boehringer Ingelheim Investigational Site, Fridley, Minnesota
  - 1311.2.10001 Boehringer Ingelheim Investigational Site, East Windsor, New Jersey
  - 1311.2.10009 Boehringer Ingelheim Investigational Site, Verona, New Jersey
  - 1311.2.10007 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1311.2.10005 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1311.2.10006 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1311.2.10011 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1311.2.10012 Boehringer Ingelheim Investigational Site, Spokane, Washington
- Canada (4):
  - 1311.2.20002 Boehringer Ingelheim Investigational Site, Markham, Ontario
  - 1311.2.20005 Boehringer Ingelheim Investigational Site, Peterborough, Ontario
  - 1311.2.20003 Boehringer Ingelheim Investigational Site, Waterloo, Ontario
  - 1311.2.20004 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- Finland (2):
  - 1311.2.35802 Boehringer Ingelheim Investigational Site, Helsinki
  - 1311.2.35801 Boehringer Ingelheim Investigational Site, Turku
- France (6):
  - 1311.2.33005 Boehringer Ingelheim Investigational Site, Marseille
  - 1311.2.33002 Boehringer Ingelheim Investigational Site, Nice
  - 1311.2.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1311.2.33004 Boehringer Ingelheim Investigational Site, Pessac
  - 1311.2.33003 Boehringer Ingelheim Investigational Site, Rouen
  - 1311.2.33006 Boehringer Ingelheim Investigational Site, Toulouse
- Germany (5):
  - 1311.2.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1311.2.49003 Boehringer Ingelheim Investigational Site, Dresden
  - 1311.2.49005 Boehringer Ingelheim Investigational Site, Lübeck
  - 1311.2.49002 Boehringer Ingelheim Investigational Site, Mainz
  - 1311.2.49004 Boehringer Ingelheim Investigational Site, Münster
- Norway (2):
  - 1311.2.47002 Boehringer Ingelheim Investigational Site, Ålesund
  - 1311.2.47001 Boehringer Ingelheim Investigational Site, Oslo
- 1311.2.46001 Boehringer Ingelheim Investigational Site, Stockholm, Sweden

REFERENCES:
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118
- [Derived] Papp KA, Blauvelt A, Bukhalo M, Gooderham M, Krueger JG, Lacour JP, Menter A, Philipp S, Sofen H, Tyring S, Berner BR, Visvanathan S, Pamulapati C, Bennett N, Flack M, Scholl P, Padula SJ. Risankizumab versus Ustekinumab for Moderate-to-Severe Plaque Psoriasis. N Engl J Med. 2017 Apr 20;376(16):1551-1560. doi: 10.1056/NEJMoa1607017. PMID 28423301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow shows disposition at the end of treatment.
Groups:
- BI 655066 18 mg: 18 mg BI 655066 administered by subcutaneous injection plus two placebo matching BI 655066 injections at Week 0, followed by two placebo matching BI 655066 injections each at Weeks 4 and 16.
- BI 655066 90 mg: 90 mg BI 655066 administered by subcutaneous injection plus two placebo matching BI 655066 injections at Week 0, followed 90mg BI 655066 plus one placebo matching BI 655066 injection at Weeks 4 and 16.
- BI 655066 180 mg: 180 mg BI 655066 administered by subcutaneous injection as two injections plus a placebo matching BI 655066 injection at Week 0, followed 180 mg BI 655066 administered as two injections at Weeks 4 and 16.
- Stelara: Stelara administered by subcutaneous injection plus two saline injections at Week 0, Stelara injection plus one saline injection at Weeks 4 and 16. Stelara dose was 45 mg for patients with body weight ≤100 kg at randomisation or 90 mg for patients with body weight >100 kg at randomisation.
Period: Overall Study
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | Stelara
Started | 43 | 41 | 42 | 40
Completed | 39 | 39 | 40 | 39
Not Completed | 4 | 2 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other reason | 2 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set (SAF) which Included all randomised patients who received at least 1 dose of trial medication and was based on the first treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | Stelara | Total
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 166
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (14.2) | 49.3 (13.3) | 44.9 (14.0) | 45.4 (12.1) | 45.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 13 | 13 | 57
  Male | 23 | 30 | 29 | 27 | 109

OUTCOME MEASURES:

1. Primary Outcome: Achievement of ≥90% Reduction From Baseline PASI Score (PASI90) at Week 12
Description: Percentage of participants who achieved ≥90% reduction from baseline in Psoriasis Area and Severity Index score (PASI90) at Week 12.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) which included all randomised patients who received at least 1 dose of trial medication and was based on the randomised treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- BI 655066 90+180 mg: 90 mg BI 655066 or 180mg BI 655066 administered by subcutaneous injection at Weeks 0, 4 and 16, plus matching placebos.
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants | 32.6 [19.1 to 48.5] | 73.2 [57.1 to 85.8] | 81.0 [65.9 to 91.4] | 77.1 [66.6 to 85.6] | 40.0 [24.9 to 56.7]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for weight (=<100kg vs >100kg) & prior exposure to 2 or more tumour necrosis factor antagonists with discontinuation due to lack of efficacy; Mean Difference (Net) = 36.4, 95% CI 2-sided [19.0 to 53.8] — Difference calculated as BI 90+180 mg minus Stelara

2. Secondary Outcome: Achievement of ≥75% Reduction From Baseline in PASI Score (PASI75) at Weeks 12 and 24
Description: Percentage of participants who achieved ≥75% reduction from baseline in Psoriasis Area and Severity Index score (PASI75) at Weeks 12 and 24.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Baseline, Week 12 and Week 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants
  Week 12 | 67.4 [51.5 to 80.9] | 97.6 [87.1 to 99.9] | 90.5 [77.4 to 97.3] | 94.0 [86.5 to 98.0] | 77.5 [61.5 to 89.2]
  Week 24 | 55.8 [39.9 to 70.9] | 92.7 [80.1 to 98.5] | 92.9 [80.5 to 98.5] | 92.8 [84.9 to 97.3] | 70.0 [53.5 to 83.4]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Week 12; Test type: Superiority or Other; p = 0.0355, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 14.6, 95% CI 2-sided [1.0 to 28.2] — Difference calculated as BI 90+180 mg minus Stelara
Statistical Analysis 2: Comparison: BI 655066 90+180 mg vs Stelara; Week 24; Test type: Superiority or Other; p = 0.0062, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 21.1, 95% CI 2-sided [6.0 to 36.2] — Difference calculated as BI 90+180 mg minus Stelara

3. Secondary Outcome: Achievement of 100% Reduction From Baseline in PASI Score (PASI100) at Week 12
Description: Percentage of participants who achieved 100% reduction from baseline in Psoriasis Area and Severity Index score (PASI100) at Week 12.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Baseline and Week 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants | 14.0 [5.3 to 27.9] | 41.5 [26.3 to 57.9] | 50.0 [34.2 to 65.8] | 45.8 [34.8 to 57.1] | 17.5 [7.3 to 32.8]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 27.1, 95% CI 2-sided [11.3 to 42.9] — Difference calculated as BI 90+180 mg minus Stelara

4. Secondary Outcome: Achievement of ≥50% Reduction From Baseline in PASI Score (PASI50) at Week 12
Description: Percentage of participants who achieved ≥50% reduction from baseline in Psoriasis Area and Severity Index score (PASI50) at Week 12.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Baseline and Week 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants | 93.0 [80.9 to 98.5] | 100.0 [91.4 to 100.0] | 95.2 [83.8 to 99.4] | 97.6 [91.6 to 99.7] | 87.5 [73.2 to 95.8]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p = 0.0706, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 10.1, 95% CI 2-sided [-0.8 to 21.1] — Difference calculated as BI 90+180 mg minus Stelara

5. Secondary Outcome: Achievement of PASI90 at Week 24
Description: Percentage of participants who achieved PASI90 at Week 24.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Week 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants | 30.2 [17.2 to 46.1] | 65.9 [49.4 to 79.9] | 85.7 [71.5 to 94.6] | 75.9 [65.3 to 84.6] | 55.0 [38.5 to 70.7]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p = 0.0300, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 19.8, 95% CI 2-sided [1.9 to 37.7] — Difference calculated as BI 90+180 mg minus Stelara

6. Secondary Outcome: Percentage Change in PASI Score From Baseline at Week 12
Description: Percentage change in Psoriasis Area and Severity Index (PASI) from baseline at Week 12.
  PASI score ranges from 0 (best) to 72 (worst).
Time Frame: Baseline and Week 12
Population: FAS including patients with available data.
Measure: Mean (Standard Deviation); unit: Percentage of PASI score
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 39 | 41 | 41 | 82 | 37
Percentage of PASI score | -79.7 (19.5) | -93.4 (7.7) | -90.7 (23.1) | -92.1 (17.1) | -82.1 (19.5)

7. Secondary Outcome: Achievement of sPGA Clear or Almost Clear at Week 12
Description: Percentage of participants who achieved static Physician Global Assessment (sPGA) clear or almost clear at Week 12.
  sPGA is assessed on a six-point scale from 0 (clear) to 5 (severe).
Time Frame: Week 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Percentage of participants | 62.8 [46.7 to 77.0] | 90.2 [76.9 to 97.3] | 90.5 [77.4 to 97.3] | 90.4 [81.9 to 95.7] | 67.5 [50.9 to 81.4]
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p = 0.0072, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 21.2, 95% CI 2-sided [5.7 to 36.6] — Difference calculated as BI 90+180 mg minus Stelara

8. Secondary Outcome: Time to Loss of PASI50 Response
Description: Time to loss of PASI50 response.
Time Frame: From first drug administration until end of follow-up period, up to 48 weeks
Population: FAS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | BI 655066 90+180 mg | Stelara
Number analyzed (Participants) | 43 | 41 | 42 | 83 | 40
Days | 253 [212 to 285] | NA [NA to NA] — Not calculable due to low number of patients with events | NA [NA to NA] — Not calculable due to low number of patients with events | NA [NA to NA] — Not calculable due to low number of patients with events | 338 [253 to NA] — Not calculable due to low number of patients with events
Statistical Analysis 1: Comparison: BI 655066 90+180 mg vs Stelara; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.1844, 95% CI 2-sided [0.1 to 0.4]

ADVERSE EVENTS:
Time Frame: From first drug administration until 15 weeks after the last drug administration, up to 231 days
Arm/Group | BI 655066 18 mg | BI 655066 90 mg | BI 655066 180 mg | Stelara
Serious Adverse Events (participants affected / at risk) | 5/43 | 6/41 | 0/42 | 3/40
Other Adverse Events (participants affected / at risk) | 23/43 | 22/41 | 20/42 | 17/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655066 18 mg (N=43) | BI 655066 90 mg (N=41) | BI 655066 180 mg (N=42) | Stelara (N=40)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655066 18 mg (N=43) | BI 655066 90 mg (N=41) | BI 655066 180 mg (N=42) | Stelara (N=40)
Folliculitis (Infections and infestations) | 3 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 15 | 14 | 11 | 5
Rhinitis (Infections and infestations) | 0 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Headache (Nervous system disorders) | 5 | 2 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.